CLINICAL TRIAL: NCT05603858
Title: The Role of End Button Tenodesis in the Management of Failed Developmental Dysplasia of the Hip Surgery
Brief Title: End Button Tenodesis in Failed Developmental Dysplasia of the Hip Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Obeid Abd Allah, Principal Investigator, Al-Azhar University
Other Study IDs: EBT
Record Dates: First submitted 2022-10-29; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tenodesis by end button: open reduction of the dislocated hip and stabilization by end button
  Interventions: Procedure: Tenodesis by end button

INTERVENTIONS:
Procedure: Tenodesis by end button — open reduction of the dislocated hip and stabilization by end button

SUMMARY:
Adequate growth and development of the hip depends on two main factors: concentric positioning of femoral head into the acetabular cavity and adequate balance in growth between tri-radiate and acetabular cartilage. Any alteration in these two conditions leads to a hip dysplasia & dislocation

ELIGIBILITY:
Inclusion Criteria:

- Patient with Developmental dysplasia of the hip (DDH) with :

* Age: up to 9 years old.
* Recurrent DDH .
* Failed open reduction through medial approach in the management of DDH.
* Traumatic hip dislocation .

Exclusion Criteria:

* • Paralytic hip dislocation .

  * Post septic hip dislocation.
  * Refusal to participate in this study.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients will be examined for:
  Length of both lower limbs in relation to each other. Length of both lower limbs according to patient age. Presence of hump related to the outer surface of the hip Presence of pain, abnormal gait, Trendlenburg test Radiographic evaluation (antero posterior and frog pelvis views)
  An addition to the steps of the open reduction, the following were done:
  1. Trans articular suturing
  2. End button tenodesis
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2022-11-29 (Estimated); Primary Completion 2023-11-29 (Estimated); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
modified Harris Hip Score | 6 months
  score for function of the hip

REFERENCES:
- [Background] Zhang S, Doudoulakis KJ, Khurwal A, Sarraf KM. Developmental dysplasia of the hip. Br J Hosp Med (Lond). 2020 Jul 2;81(7):1-8. doi: 10.12968/hmed.2020.0223. Epub 2020 Jul 6. PMID 32730146
- [Background] Schaeffer EK, Study Group I, Mulpuri K. Developmental dysplasia of the hip: addressing evidence gaps with a multicentre prospective international study. Med J Aust. 2018 May 7;208(8):359-364. doi: 10.5694/mja18.00154. PMID 29716513